CLINICAL TRIAL: NCT01033617
Title: The IMPlantation of Autologous CD133+ sTem Cells in Patients Undergoing CABG With Left Ventricular Dysfunction: the IMPACT-CABG Study
Brief Title: IMPACT-CABG Trial: IMPlantation of Autologous CD133+ sTem Cells in Patients Undergoing CABG
Acronym: IMPACT-CABG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Miltenyi Biotec, Inc. (Industry); Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other); Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HD08.147
Record Dates: First submitted 2009-12-14; First posted 2009-12-16 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2015-07

CONDITIONS: Myocardial Infarct; Heart Failure
Keywords: Stem cells; Cellular therapy; Myocardial repair
MeSH Terms: conditions — Myocardial Infarction; Heart Failure

STUDY DESIGN:
Intervention Model Description: Stem cell or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Saline solution with autologous plasma.
  Interventions: Procedure: Injection of stem cells at time of coronary artery bypass grafting
- CD133+ stem cells (Experimental): Autologous CD133+ intramyocardial injection at time of coronary artery bypass grafting.
  Interventions: Procedure: Injection of stem cells at time of coronary artery bypass grafting

INTERVENTIONS:
Procedure: Injection of stem cells at time of coronary artery bypass grafting — Following completion of the distal coronary artery bypasses, autologous CD133+ stem cells,or placebo solution containing plasma and indistinguishable will be injected in the myocardium. A total of 2.0 ml with 10-15 injections will be injected.
  Other Names: CD133+ autologous stem cells OR placebo solution containing autologous plasma

SUMMARY:
Following myocardial infarct, cellular therapy is a potential approach to repopulate the injured myocardium, to treat heart failure and restore cardiac function. The purpose of this study is to assess the safety, feasibility and efficacy of intramyocardial delivery of selected autologous CD133+ bone marrow stem cells at time of coronary artery bypass grafting in patients with chronic ischemic cardiomyopathy.

DETAILED DESCRIPTION:
CD133+ are well-characterized distinct early progenitor group of stem cells that possess high engraftment, pluripotent and angiogenic capacity and proved to be valuable for cardiac repair by promoting neovascularization, inhibition of apoptosis and cardiomyogenesis.

Our proposed research protocol involves patients with chronic ischemic heart disease and left ventricular dysfunction undergoing coronary artery bypass grafting (CABG). In this phase II clinical trial, prospective, randomized, 2 arm, double-blind, placebo-controlled study, we will assess the safety, feasibility and functional effect of intra-myocardial injection of highly selected autologous CD133+ bone marrow stem cells to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, and ≤75 years.
* Patients with severe chronic ischemic cardiomyopathy manifested by Canadian Cardiovascular Society (CCS) class II or greater angina, and/or New York Heart Association (NYHA) class II or greater, AND who have undergone diagnostic coronary angiography demonstrating ≥70% diameter narrowing of at least 2 major coronary arteries or branches or ≥50% diameter narrowing of the left main coronary artery.
* A significant left ventricular systolic dysfunction evaluated by echocardiography or LV angiography (LV ejection fraction ≤45% but ≥25%) due to prior myocardial infarction. This area of left ventricular dysfunction should be akinetic or severely hypokinetic, not dyskinetic or aneurismal, when assessed by echocardiography or LV angiogram. This territory should be irrigated by one or a branch of the three major vascular territories (i.e. right coronary artery, left circumflex, or left anterior descending artery distribution) that will be bypassed during the surgical procedure.
* No contraindications or exclusions (see below).
* Willingness to participate and ability to provide informed consent.

Exclusion Criteria:

* Contraindications to magnetic resonance imaging including presence of an implantable cardiac defibrillator (ICD) or permanent pacemaker (PPM), or cases in which it is anticipated that an ICD or PPM will be implanted prior to the 6 month follow-up (thus precluding performance of follow-up MR scans), claustrophobia.
* Lack of ischemic symptoms (angina) prior to referral for CABG (i.e., patients with only 'silent' ischemia will be excluded).
* Need for urgent or emergent revascularization.
* Need for concomitant surgical procedure at the time of CABG (e.g. valve repair or replacement, aneurysm resection, etc.).
* Hemodynamically unstable patients, as defined by heart rate ≤40/min or ≥100/min, and/or systolic blood pressure <90 mmHg or ≥200 mmHg, and/or ongoing need for intravenous inotropic or vasopressor medications.
* Patients with confirmed myocardial infarction within 14 days, and/or rising cardiac biomarker proteins (i.e. troponin), and/or worsening ECG changes.
* Prior CABG surgery.
* Stroke within 3 months prior to planned CABG.
* Immunosuppressive medication (e.g. prednisone, cyclophosphamide, etanercept, etc.)
* Severe chronic renal insufficiency (serum creatinine ≥ 200 mmol/dl or need for dialysis), liver disease, (diagnosis of cirrhosis, chronic hepatitis, or elevation of serum transaminases ≥3 times the upper limit of normal), cerebrovascular disease requiring concomitant carotid endarterectomy, peripheral arterial disease (claudication as the primary factor limiting activity), active non-dermatological malignancy requiring on-going treatment, or any other condition that would place the patient at increased risk for complications in the judgment of the attending cardiologist or cardiac surgeon
* Contra-indication for bone marrow aspiration (Thrombocytopenia <50.000 mm3, INR >2.0, use of antiplatelet agents other than aspirin).
* Hemoglobin less than 10g/dL, white blood cell count less than 4,000/mm3, absolute neutrophil count less than 1500/mm3
* Active infection, with a temperature greater than 37.5°C within 48 hrs prior to surgery and an unexplained white blood cell count in excess of 10,000/mm3
* Myelodysplastic syndrome (MDS)
* Significant cognitive impairment
* Any condition associated with a life expectancy of less than 6 months
* Patients known allergic reaction or contraindication to any of the component of the CD133+ enriched cells
* Participation in other studies
* History of severe ventricular tachy-arrythmias
* Positive laboratory test results for syphilis, HIV, HBC, HCV, HTLV1 and HTLV2
* Pregnant woman
* Inability or unwillingness to provide written informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-12; Primary Completion 2014-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Freedom from Major Adverse Cardiac Event: cardiac death, myocardial infarct, repeat coronary bypass grafting or percutaneous intervention of bypassed artery. | 6 months
Freedom from major arrhythmia: sustained ventricular tachycardia or survived sudden death. | 6 months

SECONDARY OUTCOMES:
Regional myocardial perfusion and function assessed by magnetic resonance scans. | 6 months
Device performance end point: Feasibility to produce from 100ml of bone marrow aspiration a final cell product that contains a target CD133+ cells higher than 0.5 million with a purity superior to 30% and a recovery superior to 10%. | Baseline
On symptom severity and quality of life after CABG surgery. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Noiseux, MD, MSc, FRCSC, Principal Investigator — Montreal University
Locations (1):
- Centre de recherche du CHUM (CRCHUM), Montreal, Quebec, Canada

REFERENCES:
- [Derived] Noiseux N, Mansour S, Weisel R, Stevens LM, Der Sarkissian S, Tsang K, Crean AM, Larose E, Li SH, Wintersperger B, Vu MQ, Prieto I, Li RK, Roy DC, Yau TM. The IMPACT-CABG trial: A multicenter, randomized clinical trial of CD133+ stem cell therapy during coronary artery bypass grafting for ischemic cardiomyopathy. J Thorac Cardiovasc Surg. 2016 Dec;152(6):1582-1588.e2. doi: 10.1016/j.jtcvs.2016.07.067. Epub 2016 Aug 13. PMID 27665225